CLINICAL TRIAL: NCT05780749
Title: A 14-week Pilot Prospective Clinical Trial With BiOkuris Product in Patients With Irritable Bowel Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biokuris s.a. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: BK-IBS-2301
Record Dates: First submitted 2023-03-09; First posted 2023-03-23 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS; chitin-glucan
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, double-blind, placebo controlled, multicenter, parallel group study. Patients will be recruited in multiple centers in Belgium.
  Patients will be treated for a total of 12 weeks. The study consists of a 2 weeks run-in period followed by a 8 weeks treatment period with DDI-IBS-001. At the end of the 8 weeks treatment, patients will be divided in responders and non-responders based on their global symptoms' relief score (patients will be considered responders with a weekly SGA score mean of 3 points or less for at least 50% of the 6 last weeks of treatment before week 10 [week 4 to 10]).
  Responder patients will be randomised in a 2:1 allocation ratio to receive either DDI-IBS-001 or placebo, for 4 additional weeks. Non-responder patients will continue the treatment with DDI-IBS-001 for additional 4 weeks. The study period will be followed by a follow-up period of 4 weeks during which patients will have free access to DDI-IBS-001.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The stage 2 of this study is a double-blinded study. Neither patients, nor investigators, nor trial staff, nor the sponsor study team will be aware of treatment assignments prior to the database lock at the conclusion of the study. The study products are DDI-IBS-001 and its matching placebo. DDI-IBS-001 and placebo will be provided as sachets containing 1980mg of powder to be dissolved in a glass of water (about 250 ml) and taken orally, with the same composition except for the active ingredient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active arm - DDI-IBS-001 (Experimental)
  Interventions: Dietary Supplement: DDI-IBS-001
- Placebo arm (Placebo Comparator)
  Interventions: Other: DDDI-IBS-001 placebo

INTERVENTIONS:
Dietary Supplement: DDI-IBS-001 — The product is a combination of chitin-glucan and other dietary complement components. The dosage of chitin-glucan is 1.5 g/day. The product is a powder for oral administration 1x/day.
  Arms: Active arm - DDI-IBS-001
Other: DDDI-IBS-001 placebo — The placebo product has the same composition in excipient, same form and same posology as DDI-IBS-001.
  Arms: Placebo arm

SUMMARY:
Irritable Bowel Syndrome (IBS) is a common chronic gastrointestinal condition that affects approximately 10-20% of adults in Western countries. IBS is a disorder with chronic or recurrent colonic symptoms without a clear-cut etiology. This condition is characterized by chronic or recurrent ABDOMINAL PAIN, bloating, MUCUS in FECES, and an erratic disturbance of DEFECATION. Symptoms include cramping, abdominal pain, bloating, gas, and diarrhea or constipation, or both. Over 80% of individuals with IBS report food-related symptoms leading in the 70% of these patients to self-imposed food restrictions and/or modifications of their diet. These spontaneous unsupervised dietary modifications are associated with maladaptive eating patterns and unnecessary self-restricted diets, which could result in nutritional deficiencies.

BiOkuris product DDI-IBS-001 is a food multicomponents product based on BiOkuris proprietary chitin-glucan complex. The objectives of the VITABIOTIC study is to confirm the effectiveness of the DDI-IBS-001 product in improving global symptoms, abdominal pain, stool consistency, quality of life, anxiety and depression in IBS patients and to confirm the product's safety.

ELIGIBILITY:
Inclusion Criteria:

1. Adult females and males, aged 18-75 years,
2. Diagnosis of IBS at least 6 months prior to study entry,
3. Confirmed IBS according to Rome-IV criteria (as determined by investigator),
4. Patient having either constipation (IBS-C), diarrhoea (IBS-D) or alternance of constipation/diarrhoea (IBS-M),
5. Possession of a digital device (i.e., smartphone or tablet),
6. Patient who read, understood, and signed the informed consent form (ICF),
7. Patient willing to adhere to the study visit schedule and capable to understand and comply with protocol requirements and product intake,
8. Male, or female patient of childbearing potential, who agrees to use acceptable birth control methods throughout the study period.

   As assessed at the end of the run-in period, week 2 :
9. Patient with a baseline score for abdominal pain ≥ 2 and < 6 assessed on a 7-point Lickert scale
10. Patient with correct and complete reporting of the study questionnaires and scores during the run-in period (≥75% completion)

Exclusion Criteria:

1. Severe gastrointestinal pathologies other than IBS, including: ulcers, coeliac disease, inflammatory bowel disease, bowel cancer, bowel resection, auto-immune diseases (e.g., rheumatoid arthritis, systemic lupus erythematosus, multiple sclerosis, Graves' disease), bariatric surgery, acute or chronic diarrhoea secondary to confirmed infectious gastroenteritis, or enteral or parenteral nutrition,
2. Metabolic disorders affecting intestinal transit function or nutrient absorption including uncontrolled diabetes and uncontrolled dysthyroidism,
3. Patients experiencing complications of abdominal radiotherapy,
4. Surgical operations to the mouth or gastrointestinal tract within 4 weeks prior to study entry, or planned during the study; appendectomy within 6 months prior to study entry,
5. Galactose intolerance ,
6. Use of opioids or narcotic analgesics within 6 weeks prior to week 0,
7. Systemic antibiotic treatment in progress or prescribed less than 4 weeks prior to study entry,
8. Use of products marketed as or rich in prebiotics, probiotics, or symbiotics (e.g., kefir, probiotic yogurt, baker's yeast, etc.) less than 2 weeks prior to week 0,
9. Use of laxatives, antibloating agents, antidiarrheal medication, antispasmodics, anxiolytics, antidepressants, analgesics, and non-steroidals anti-inflammatory drugs if started less than 2 months prior to week 0 . These medications are authorized if consumed for longer than 2 months before week 0 and maintained at a stable dosage for the entire study duration,,
10. Diets including low-FODMAP, KETO/high-fat, gluten free/coeliac, paleo, weight loss, caloric restriction, low-carb, 5:2/whole day energy restriction, Atkins/high-protein, sugar-free, single-food, juicing/any day of juicing, any other restriction diet (e.g. very low calory), or vegan diets if started less than 2 months prior or stopped less than 1 month prior to week 0. These diets are authorized if followed for longer than 2 months before week 0 and maintained for the entire study duration,,
11. Excessive alcohol consumption (more than 10 units per week) and/or drug abuse,
12. Pregnancy and lactation, or plan to become pregnant during the study period,
13. Participation in other studies involving investigational or marketed products concomitantly or less than 3 months prior to study entry,
14. Known hypersensitivity to any of the ingredients or excipients of the investigational products,
15. Patient who has forfeited their freedom by administrative or legal award, or who is under guardianship or under limited judicial protection.

    As assessed at the end of the run-in period, week 2 :
16. Use of opioids or narcotic analgesics during the run-in period (between week 0 and week 1),
17. Systemic antibiotic treatment in progress or prescribed during the run-in period (between week 0 and week 1),
18. Deviation from lifestyle and dietary recommendations to be followed during the study (between week 0 and week 1).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2023-11-23 (Actual); Primary Completion 2025-02-02 (Actual); Study Completion 2025-02-02 (Actual)

PRIMARY OUTCOMES:
Symptoms global assessment of relief (SGA) responder rate | Week 10 (8 weeks after run-in period)
  The primary outcome is the subjective global assessment (SGA) of relief responder rate at Week 8. Patients with an SGA of relief score of 3 points or less each week will be considered weekly responders. Patients who respond weekly for at least 50% of assessments after 2 weeks of Biokuris food supplement administration until V3 will be considered overall responders.

SECONDARY OUTCOMES:
Weekly SGA responder rate | weekly from week 2 to week 14
  The SGA of relief weekly responder rate after 8 weeks of Biokuris food supplement administration. Patients with an SGA of relief score of 3 points or less each week will be considered weekly responders.
Individual symptoms | weekly from week 2 to week 14
  Weekly change from baseline in mean 7-point Likert scale for each of the symptoms: abdominal pain, abdominal bloating, flatulence, dyschezia, pain during evacuation. Patients will score the intensity of each symptom individually from 1 (none) to 7 (very severe). Incidence of responders.
stool consistency | weekly from week 2 to week 14
  Change in the weekly mean number of normal stool consistency, evaluated with the BSS. Stool consistency (BSS score) will be described for each week until V4. The change in the weekly average number of normal stool consistency will be calculated between week 2 (baseline), and each week of treatment
number of evacuation per day | weekly from week 2 to week 14
  Change in the weekly mean number of evacuations per day. The mean daily number of bowel movements will be calculated for each week until week 14. The change in the weekly average number of evacuations will be calculated between week 2 (baseline), and each week of treatment, until week 14. A stratification will be performed according to weekly mean numbers registered at week 2.
IBS-QoL | Week 0, week 4, week 8, week 10, week 14
  Absolute and relative change of IBS-QoL (Quality of Life) score. An analysis for each of the 8 domains of the validated questionnaire will be performed.
Anxiety & Depression | Week 0, week 4, week 8, week 10, week 14
  Monthly change from baseline in Hospitalization Anxiety and Depression Scale (HADS) score. It is divided into an anxiety subscale (HADS-A) and a depression subscale (HADS-D), both containing 7 intermingled items, and are scored separately. For both scales, scores of less than 7 indicate non-cases, and between 8-10 mild, 11-14 moderate and 15-21 severe symptomatology.
Adverse events | Week 0, week 2, week 4, week 8, week 10, week 14
  occurrence and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, Professor, Principal Investigator — UZ Leuven
Locations (11):
- Belgium (11):
  - Centre Hospitalier EpiCURA, Ath
  - AZ Sint-Jan, Bruges
  - AZ Sint-Lucas, Bruges
  - CUB Hôpital Erasme, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - AZ Sint-Lucas, Ghent
  - UZ Brussel, Jette
  - UZ Leuven, Leuven
  - CHU Liege, Liège
  - Clinique CHC Mont-Legia, Liège
  - Centre Hospitalier du Bois de l'Abbaye, Seraing

IPD SHARING:
Plan to Share IPD: No